CLINICAL TRIAL: NCT02377830
Title: CYCLE Pilot: A Pilot Randomized Study of Early Cycle Ergometry Versus Routine Physiotherapy in Mechanically Ventilated Patients
Brief Title: CYCLE Pilot Randomized Trial
Acronym: CYCLE Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Hamilton Health Sciences Corporation (Other); Technology Evaluation in the Elderly Network / Canadian Frailty Network (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Lung Association (Other); Canadian Respiratory Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIREB 14-531
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Care; Mechanical Ventilation; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Cycling and routine physiotherapy (Experimental): Patients will receive 30 minutes of in-bed cycling in addition to routine physiotherapy, 5 days per week, for the duration of their ICU stay
  Interventions: Device: In-bed cycle ergometer (Restorative Therapies RT300 Supine)
- Routine physiotherapy (Active Comparator): Patients will receive routine physiotherapy per current institutional practice
  Interventions: Other: Routine physiotherapy

INTERVENTIONS:
Device: In-bed cycle ergometer (Restorative Therapies RT300 Supine)
  Other Names: Restorative Therapies RT300 Supine
  Arms: Early Cycling and routine physiotherapy
Other: Routine physiotherapy — activities to assist with optimizing airway clearance and respiratory function, and, based on the patient's alertness and medical stability, activities to maintain or increase limb range of motion and strength, in- and out of bed mobility, and ambulation
  Arms: Routine physiotherapy

SUMMARY:
Background: Patients in the intensive care unit (ICU) are the sickest in hospital, and need advanced life-support. Survivors of critical illness are very weak and disabled. Up to 1 in 4 have severe leg weakness impairing their quality of life for as long as 5 years after ICU discharge. In-bed cycling involves use of special equipment that attaches to a patient's hospital bed, allowing them gentle exercise while in the ICU.

Methods: Adult patients admitted to the ICU who need a breathing machine and are expected to survive their ICU stay are eligible. Patients will randomly receive 30 minutes of in-bed cycling each day they are in the ICU or routine physiotherapy, both delivered by specially trained physiotherapists.

Outcomes: Feasibility: The investigators will study whether patients can cycle on most days of their ICU stay, whether patients and their families agree to be a part of the study, and whether investigators can systematically assess patients' strength.

Relevance: Effective methods of physiotherapy are needed for critically ill patients to minimize muscle weakness, speed recovery, and improve quality of life. This pilot randomized study is the second of several future larger studies about in-bed cycling in the ICU.

Our pilot work includes CYCLE Pilot and CYCLE Vanguard. CYCLE Pilot is an external pilot and enrolled 66 patients from 3/2015 to 6/2016. CYCLE Vanguard is an internal pilot and enrolled 47 patients from 11/2016 to 3/2018. CYCLE Vanguard patients will be analyzed in the main CYCLE RCT (NCT03471247).

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to a medical-surgical ICU within the 1st 4 days of mechanical ventilation (MV) and 1st 7 days of ICU, and
* could ambulate independently before hospital admission.

Exclusion Criteria:

* Acute condition impairing patients' ability to cycle (e.g., leg fracture),
* proven or suspected neuromuscular weakness affecting the legs (e.g., stroke or Guillain-Barré syndrome),
* unable to follow commands in English pre-ICU,
* temporary pacemaker,
* expected hospital mortality >90%,
* unable to fit the bike, palliative goals of care, or persistent therapy exemptions in the 1st 4 days of MV (e.g., cardiorespiratory instability, active major bleeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient accrual | 2 years

SECONDARY OUTCOMES:
Cycling protocol violations (% cycling protocol violations) | 2 years
  % cycling protocol violations
Outcome measure ascertainment (% outcomes measured in hospital) | 2 years
  % outcomes measured in hospital
Blinded outcome measures at hospital discharge (% outcomes at hospital discharge measured by blinded outcome assessors) | 2 years
  % outcomes at hospital discharge measured by blinded outcome assessors
Physical Function Test for ICU (PFIT) at ICU awakening, ICU discharge, 3-days post-ICU discharge (CYCLE Vanguard only) and hospital discharge | From study admission to approximately 5, 12, 15 and 30 days, on average, respectively
  Patients complete 4 activities: arm and leg strength, ability to stand, and step cadence. Scores range from 0 to 10, with higher scores = better function
Muscle strength at ICU awakening, ICU discharge, 3-days post-ICU discharge (CYCLE Vanguard only), and hospital discharge | From study admission to approximately 5, 12, 15 and 30 days, on average, respectively
  Manual muscle testing using the Medical Research Council (MRC) Scale. The patient exerts a force against the examiner's resistance. Each muscle is assessed on a 6-point MRC scale (0=no contraction; 5=contraction sustained against maximal resistance).
Quadriceps strength at ICU and hospital discharge (Force measured in Kg and in Newtons on a continuous scale) | From study admission to approximately 12 and 30 days, on average, respectively
  The patient exerts a force against a small strain gauge that fits in the examiner's hand. .
2 minute walk test at ICU discharge, 3-days post-ICU (CYCLE Vanguard only), and hospital discharge | From study admission to approximately 12 and 30 days, on average, respectively
  Maximum distance walked in 2 minutes measured in metres on a continuous scale

OTHER OUTCOMES:
Katz Activities of Daily Living Scale at ICU and hospital discharge | From study admission to approximately 12 and 30 days, on average, respectively
  The patient's ability to complete 6 tasks: bathing, dressing, toileting, feeding, continence, and bed mobility. A rater assesses whether the patient is dependent or independent according to pre-specified criteria.
Euro-QOL 5DL | From study admission to approximately 12 and 30 days, on average, respectively
  5 question self-administered, preference-based instrument to measure mobility, self-care, usual activities, pain, and anxiety/ depression, as well as a global assessment of health

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kho, PT, PhD, Principal Investigator — McMaster University School of Rehabilitation Science
Locations (9):
- Duke University Medical Center, Durham, North Carolina, United States
- Austin Health, Melbourne, Victoria, Australia
- Canada (7):
  - St. Joseph's Healthcare Intensive Care Unit, Hamilton, Ontario
  - Hamilton Health Sciences General ICU, Hamilton, Ontario
  - Hamilton Health Sciences Juravinski ICU, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Kho ME, Molloy AJ, Clarke FJ, Reid JC, Herridge MS, Karachi T, Rochwerg B, Fox-Robichaud AE, Seely AJ, Mathur S, Lo V, Burns KE, Ball IM, Pellizzari JR, Tarride JE, Rudkowski JC, Koo K, Heels-Ansdell D, Cook DJ. Multicentre pilot randomised clinical trial of early in-bed cycle ergometry with ventilated patients. BMJ Open Respir Res. 2019 Feb 18;6(1):e000383. doi: 10.1136/bmjresp-2018-000383. eCollection 2019. PMID 30956804
- [Derived] Heels-Ansdell D, Kelly L, O'Grady HK, Farley C, Reid JC, Berney S, Pastva AM, Burns KE, D'Aragon F, Herridge MS, Seely A, Rudkowski J, Rochwerg B, Fox-Robichaud A, Ball I, Lamontagne F, Duan EH, Tsang J, Archambault PM, Verceles AC, Muscedere J, Mehta S, English SW, Karachi T, Serri K, Reeve B, Thabane L, Cook D, Kho ME. Early In-Bed Cycle Ergometry With Critically Ill, Mechanically Ventilated Patients: Statistical Analysis Plan for CYCLE (Critical Care Cycling to Improve Lower Extremity Strength), an International, Multicenter, Randomized Clinical Trial. JMIR Res Protoc. 2024 Oct 28;13:e54451. doi: 10.2196/54451. PMID 39467285
- [Derived] O'Grady HK, Ball I, Berney S, Burns KEA, Cook DJ, Fox-Robichaud A, Herridge MS, Karachi T, Mathur S, Reid JC, Rochwerg B, Rollinson T, Rudkowski JC, Bosch J, Turkstra LS, Kho ME. Characterizing usual-care physical rehabilitation in Canadian intensive care unit patients: a secondary analysis of the Canadian multicentre Critical Care Cycling to Improve Lower Extremity Strength pilot randomized controlled trial. Can J Anaesth. 2024 Oct;71(10):1406-1416. doi: 10.1007/s12630-024-02838-7. Epub 2024 Sep 24. PMID 39317833
- [Derived] Kho ME, Berney S, Pastva AM, Kelly L, Reid JC, Burns KEA, Seely AJ, D'Aragon F, Rochwerg B, Ball I, Fox-Robichaud AE, Karachi T, Lamontagne F, Archambault PM, Tsang JL, Duan EH, Muscedere J, Verceles AC, Serri K, English SW, Reeve BK, Mehta S, Rudkowski JC, Heels-Ansdell D, O'Grady HK, Strong G, Obrovac K, Ajami D, Camposilvan L, Tarride JE, Thabane L, Herridge MS, Cook DJ. Early In-Bed Cycle Ergometry in Mechanically Ventilated Patients. NEJM Evid. 2024 Jul;3(7):EVIDoa2400137. doi: 10.1056/EVIDoa2400137. Epub 2024 Jun 12. PMID 38865147
- [Derived] Kho ME, Reid J, Molloy AJ, Herridge MS, Seely AJ, Rudkowski JC, Buckingham L, Heels-Ansdell D, Karachi T, Fox-Robichaud A, Ball IM, Burns KEA, Pellizzari JR, Farley C, Berney S, Pastva AM, Rochwerg B, D'Aragon F, Lamontagne F, Duan EH, Tsang JLY, Archambault P, English SW, Muscedere J, Serri K, Tarride JE, Mehta S, Verceles AC, Reeve B, O'Grady H, Kelly L, Strong G, Hurd AH, Thabane L, Cook DJ; CYCLE Investigators and the Canadian Critical Care Trials Group. Critical Care Cycling to Improve Lower Extremity Strength (CYCLE): protocol for an international, multicentre randomised clinical trial of early in-bed cycling for mechanically ventilated patients. BMJ Open. 2023 Jun 23;13(6):e075685. doi: 10.1136/bmjopen-2023-075685. PMID 37355270
- [Derived] Takaoka A, Heels-Ansdell D, Cook DJ, Kho ME. The Association between Frailty and Short-Term Outcomes in an Intensive Care Unit Rehabilitation Trial: An Exploratory Analysis. J Frailty Aging. 2021;10(1):49-55. doi: 10.14283/jfa.2020.52. PMID 33331622
- [Derived] Reid JC, McCaskell DS, Kho ME. Therapist perceptions of a rehabilitation research study in the intensive care unit: a trinational survey assessing barriers and facilitators to implementing the CYCLE pilot randomized clinical trial. Pilot Feasibility Stud. 2019 Nov 12;5:131. doi: 10.1186/s40814-019-0509-3. eCollection 2019. PMID 31741746
- [Derived] McCaskell DS, Molloy AJ, Childerhose L, Costigan FA, Reid JC, McCaughan M, Clarke F, Cook DJ, Rudkowski JC, Farley C, Karachi T, Rochwerg B, Newman A, Fox-Robichaud A, Herridge MS, Lo V, Feltracco D, Burns KE, Porteous R, Seely AJE, Ball IM, Seczek A, Kho ME. Project management lessons learned from the multicentre CYCLE pilot randomized controlled trial. Trials. 2019 Aug 28;20(1):532. doi: 10.1186/s13063-019-3634-7. PMID 31455384
- [Derived] Kho ME, Molloy AJ, Clarke F, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Pellizzari JR, Tarride JE, Mourtzakis M, Karachi T, Cook DJ; Canadian Critical Care Trials Group. CYCLE pilot: a protocol for a pilot randomised study of early cycle ergometry versus routine physiotherapy in mechanically ventilated patients. BMJ Open. 2016 Apr 8;6(4):e011659. doi: 10.1136/bmjopen-2016-011659. PMID 27059469